CLINICAL TRIAL: NCT06160167
Title: Incidence of Hyperpigmentation in Black Patients With Multiple Myeloma Treated With Immunomodulatory Drugs
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA078-1007
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with MM treated with IMiDs
  Interventions: Drug: IMiD treatment
- Participants with MM not treated with IMiDs
  Interventions: Drug: No IMiD treatment
- Participants with MM treated with systemic therapy
  Interventions: Drug: Systemic therapy

INTERVENTIONS:
Drug: IMiD treatment — Participants with MM treated with IMiDs
  Groups: Participants with MM treated with IMiDs
Drug: No IMiD treatment — Participants with MM not treated with IMiDs
  Groups: Participants with MM not treated with IMiDs
Drug: Systemic therapy — Participants with MM treated with systemic therapy
  Groups: Participants with MM treated with systemic therapy

SUMMARY:
The purpose of this study is to measure the incidence of hyperpigmentation in Black participants with multiple myeloma (MM) treated with immunomodulatory drugs (IMiDs) compared with Black participants with MM not treated with IMiDs. The study will use de-identified data from electronic medical records in the Flatiron Health database.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age at index date
* Participants with new diagnosis of MM as defined by:

  * ICD-9-CM: 203.0x and/or ICD-10-CM: C90.0x or C90 during the study period
  * At least two documented clinical visits for MM on different days and occurring on or after January 1, 2011
* Participants who received at least one systemic MM therapy on or after initial MM diagnosis
* Participants who did not receive clinical study drug at any time during the observation period
* Participants with race information

Exclusion Criteria:

* Exclusion Criteria
* Patients with less than 6 months of medical data during the prior or follow-up period
* Patients in more than one race category (mix race), missing race, unknown race, and "other" race
* Patients diagnosed with the following hematological cancers on or prior to the index date:

  * myelodysplastic syndromes (ICD-9: 238.74, 238.75; ICD-10: D46.xx)
  * mantle cell lymphoma (ICD-9: 200.4x, ICD-10: C83.1x)
  * follicular lymphoma (ICD-9: 202.0x, ICD-10: C82.xx)
  * marginal zone lymphoma (ICD-9: 200.3x, ICD-10: C83.4x)
* Patients with evidence of skin hyperpigmentation (ICD-9: 709.00, 709.09; ICD-10: L81.0, L81.1, L81.4, L81.8) on or prior to the index date

  * 709.00 Dyschromia, unspecified
  * 709.09 Other dyschromia
  * L81.0 Post inflammatory hyperpigmentation
  * L81.1 Chloasma/melasma
  * L81.4 Other melanin hyperpigmentation
  * L81.8 Other specified disorders of pigmentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Black and non-Black participants with MM
Sampling Method: Non-Probability Sample
Enrollment: 4204 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperpigmentation in Black participants exposed to IMiDs to non-IMiDs for MM | 12 months
  Each qualified patient must have at least 6 months of medical data recorded in the Flatiron database before the index date (pre-index period) and 6 months of available data on and after the index date (follow-up period).

SECONDARY OUTCOMES:
Incidence of skin hyperpigmentation in Black, non-Black and all participants who received systemic treatment for MM | 12 months
  Each qualified patient must have at least 6 months of medical data recorded in the Flatiron database before the index date (pre-index period) and 6 months of available data on and after the index date (follow-up period).
Risk of skin hyperpigmentation in Black and non-Black participants diagnosed with MM and exposed to IMiDs | 12 months
  Each qualified patient must have at least 6 months of medical data recorded in the Flatiron database before the index date (pre-index period) and 6 months of available data on and after the index date (follow-up period).
Risk of skin hyperpigmentation in non-Black participants exposed to IMiDs versus non-IMiDs for MM | 12 months
  Each qualified patient must have at least 6 months of medical data recorded in the Flatiron database before the index date (pre-index period) and 6 months of available data on and after the index date (follow-up period).

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers-Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Flatiron Health Oncology Database, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts